CLINICAL TRIAL: NCT02942537
Title: Single Blinded Randomized Study of Volume Reduction of Uterine Fibroids After Uterine Artery Embolization Versus Computer Tomography or Ultrasound Guided Percutaneous Microwave Ablation Evaluated by Magnetic Resonance Imaging
Brief Title: Study of Volume Reduction of Uterine Fibroids After Embolization or Microwave Treatment
Acronym: MYOMIC1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Senior consultant, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYOMIC1
Record Dates: First submitted 2016-10-15; First posted 2016-10-24 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Artery Embolization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Microwave treatment
  Interventions: Device: Microwave treatment
- Control (Active Comparator): Uterine artery embolization
  Interventions: Procedure: uterine artery embolization

INTERVENTIONS:
Device: Microwave treatment — Percutaneous or vaginal application of microwave antenna with microwave treatment of fibroma
  Arms: Intervention
Procedure: uterine artery embolization — Percutaneous applicaiton of a catheter into the femoral artery and embolization of uterine artery or branches thereof
  Arms: Control

SUMMARY:
Uterine fibroids are benign tumors that occur most commonly in women of reproductive age. Symptoms of uterine fibroids may be heavy menstrual bleeding which may lead to anemia, pressure symptoms, bowel symptoms or urinary urgency. In recent years, increasing attention has been paid to the study of minimally invasive methods for treatment. Microwave ablation of myomas and endometrium has been shown to have good effect and acceptability has been high. This study aims to compare the effectiveness, feasibility and acceptability of percutaneous or per vaginal microwave ablation and uterine artery embolization for the treatment of uterine myomas in a randomized single blind study.

Primary outcome

1. Volume reduction 6 months post treatment (+/- 15 days) compared to pre treatment measured as mean volume reduction of the 3 largest fibroids evaluated by magnetic

Power calculation

To be able to show a difference between the groups in myoma shrinkage at 6 months of 75% in microwave ablation and 50%[11] in the embolization group with a standard deviation of 25% with a alpha of 0.05 and a power of 80% we would need 16 women in each group and thus need to randomize 32 women.

In order to compensate for loss to follow-up or drop out a total of 36 women will be randomized.

Patients and investigators will not be blinded. The MRI will be performed and evaluated by a blinded radiologist.

After having signed informed consent but before randomization patients will undergo MRI of the uterine fibroids. Patients with a single fibroid measuring more than mean diameter 8cm will be excluded from further participation in the study.

All women included in the study after MRI examination will fill in a PBAC evaluation[7] during the menses preceding treatment. Women will fill a VAS for maximal pain during 1 month prior to treatment.

Microwave ablation will be performed percutaneously or vaginally using a Covidien Emprint microwave ablation system. Embolization will be performed in conscious women with an epidural catheter for pain relief.

At follow up visit 1, 3 months and 6 months post treatment acceptability will be assessed as overall satisfaction of treatment on a scale from 1-7 and if the woman would recommend the treatment to a friend.

A new MRI scan will be performed 6 months post treatment (+/-15 days).

DETAILED DESCRIPTION:
Background

Uterine fibroids are benign tumors that occur most commonly in women of reproductive age. Symptoms of uterine fibroids may be heavy menstrual bleeding which may lead to anemia, pressure symptoms, bowel symptoms or urinary urgency. Hysterectomy remains the reference standard in the treatment of uterine fibroids. However, it may cause long-term side effects such as pain and genitovaginal prolapse. It also carries a substantial risk of short term complications such as infections and organ damage. Myomectomy is another conventional treatment, but it is associated with a recurrence rate as high as 20% according to literature. It carries the same short term risks of complications as hysterectomy but at a lower frequency.

In recent years, increasing attention has been paid to the study of minimally invasive or non-invasive therapies with uterine preservation such as uterine arterial embolization (UAE), radiofrequency (RF), microwave treatment and high intensity focused ultrasound (HIFU). RF ablation often requires the aid of a laparoscopic procedure, which is invasive. HIFU is effective in small myomas, but can be time consuming in large myomas with treatments for several hours. Ultrasound or computer tomography guided percutaneous microwave thermal ablation is minimally invasive, has low time requirements, is easy to perform, and has been broadly used for the treatment of solid tumours in organs other than the uterus with favourable effects.

Microwave ablation of myomas and endometrium has been performed in China and Japan. The effect and acceptability has been high. The research team in this study has been to China to study the treatment. We have visited the clinic and studied the procedure as well as talked to patients pre- and post operatively . The equipment at Danderyd Hospital has the same output effects as the equipment in China. Danderyd Hospital as approved the method for use in uterine myomas. However, no randomized comparative study of other minimally invasive methods has been performed.

This study aims to compare the effectiveness, feasibility and acceptability of percutaneous CT- or ultrasound guided microwave ablation and uterine artery embolization for the treatment of uterine myomas in a randomized single blind study.

Power calculation

To be able to show a difference between the groups in myoma shrinkage at 6 months of 75% in microwave ablation and 50% in the embolization group with a standard deviation of 25% with a alpha of 0.05 and a power of 80% we would need 16 women in each group and thus need to randomize 32 women.

In order to compensate for loss to follow-up or drop out a total of 36 women will be randomized.

Recruitment and Randomization

Women fulfilling inclusion criteria and without exclusion criteria will be identified at the outpatient clinic of Danderyds Hospital. Advertisement may be placed in local newspapers or on social media (Facebook and Instagram) and relevant webpages or in gynecological clinics.

Women will be randomized after having been informed orally and in written and after having signed informed consent and after fulfilling inclusion and exclusion criteria after MRI-examination. Randomization will be in random permuted blocks of 6 at a ratio of 1:1. The randomization will be according to a computer generated randomization sequence. After patients have signed informed consent and fulfill inclusion without exclusion criteria after the initial magnetic resonance imaging they will be allocated to an intervention by consecutive opening of sealed opaque envelopes containing the randomization code.

Blinding

Patients and investigators will not be blinded. The MRI will be performed and evaluated by a blinded radiologist.

Method

Pre randomization evaluation

After having signed informed consent but before randomization patients will undergo MRI of the uterine fibroids. Patients with a single fibroid measuring more than 6cm will be excluded from further participation in the study.

All women included in the study after MRI examination will fill in a PBAC evaluation during the menses preceding treatment. Women will fill a VAS for maximal pain during 1 month prior to treatment. In addition a full blood panel will be evaluated.

As for uterine artery embolization no pathologist report will be performed before any treatment.

Microwave ablation

Microwave ablation will be performed percutaneously using a Covidien Emprint microwave ablation system with a 30-90 Watts effect in 14-16 gauge needle with a ceramic tip using computer tomography with fusion technique or ultrasound for myoma imaging and needle guidance. After identification of the needle path with CT or peroperative ultrasound local anaesthesia (carbocain 1% with 0,05mg/ml adrenaline) will be given along the needle path and a small skin incision using a scalpel will made for the needle entry. Patients will be given intravenous anesthesia with spontaneous breathing or general anesthesia during treatment to minimize movement during ablation.

Uterine artery embolization

Embolization will be performed in conscious women with an epidural catheter for pain relief. A catheter will be inserted in the femoral artery to access the uterine artery during x-ray monitoring and during administration of contrast to visualize the fibroma and its supporting arterial supply. When the supporting arterial branch has been identified polyvinyl alcohol particles are released into the bloodstream. These particles cause a thrombosis in the vessel.

Evaluation post treatment

Women will estimate VAS maximum postoperative pain day of surgery and the following 7 days. In addition they will note how many days passed before all pain subsided, use of pain medication will be noted and period until resuming normal daily activities. The period of hospitalization will be noted. Menstrual blood loss (PBAC) will be noted the first menstruation, menstruation number 3 and 5 post treatment. PBAC is a validated instrument for menstrual blood loss quantification.

Follow-up visits will be after first menstruation at approximately 1 month and at 3 and 6-7 months post-treatment.

At follow up visit 1, 3 months and 6 months post treatment acceptability will be assessed as overall satisfaction of treatment on a scale from 1-7 and if the woman would recommend the treatment to a friend.

A new MRI scan will be performed 6 months post treatment (+/-15 days). Women will then be asked to participate in a long-term follow up with evaluation of fibroma growth using ultrasound and recurrence of symptoms using PBAC yearly until retraction of consent.

Clinicial significance

Uterine myomas are a benign disease but have a significant impact on the lives of women. As many as 70% of women have myomas. However, the self-reported frequency of uterine myomas differs between countries and ranges from 4% to 15% in some countries- probably depending on the use of ultrasound in gynecological practice and the information given to women. Women with self reported uterine myomas are much more likely to report on symptoms which are known to be caused by myomas such as heavy menstrual bleeding, pressure symptoms, urinary urgency and pain (dysmenhorrea and dyspareunia). Myomas remain the leading cause of hysterectomies in most western countries. As hysterectomy is a highly invasive procedure with cost for women in terms of absence from work and short and long term complications, finding new minimally invasive treatments should remain a focus of health care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 30-55 with symptomatic fibromas (pressure, heaviness, bleeding, urgency)
* Premenopausal
* Fibromas with a maximum mean diameter of cm evaluated by trans vaginal or abdominal ultrasound
* Willing to comply with protocol

Exclusion Criteria:

* Current or future childwish
* Body Mass Index >35
* Treatment with anticoagulant
* Bleeding disorder which leads to increased risk of bleeding
* Patients with single fibroid more than 6cm mean diameter according to MRI.
* Contraindication for UAE or general anesthesia

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Fibroma Volume reduction 6 months post treatment | 6 months post treatment (+/-15 days)
  Volume reduction 6 months post treatment (+/- 15 days) compared to pre treatment measured as mean volume reduction of the 3 largest fibroids evaluated by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Pain | 1-7 days post treatment
  Pain (measures as visual analogue scale, VAS)- maximum postoperative pain day of surgery and following 7 days)
Symptoms of uterine fibroids | pre-treatment-6 months post treatment
  Reduction of symptoms as pressure, urgency and coital pain, score in UFS-QoL questionnaire
Use of pain medication | pre-treatment to 6 months post treatment
  Generic drug name, number of milligrams consumed
Period of sick leave | post treament to one year
  time away from work after treatment in both groups
Period of hospitalization | post treatment to one year
  number of days
Acceptability | at 3 months and 6 months
  measure as preferred method
Days of menstrual bleeding | pre and post treatment at 3 months and 6 months
  number of days of menstrual bleeding divided into fresh bleeding and spotting
Menstrual blood loss | pre and post treatment at 3 and 6 months
  Menstrual blood loss score evaluated by the validated Pictorial Bleeding assessment chart
Quality of lite | pre and post treatment at 3 and 6 months
  Quality of life evaluated by score in the validated questionnaire Uterine Fibroid Symptoms. Quality of Life (UFS-QoL)
Complications | at any time after enrollment up to 6 months post treatment
  Any complication occurring in women will be recorded and judged by the principal investigator as related, probably related, probably not related or not related

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp Kallner, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of Obstetrics and Gynecology, Dnderyds Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Kanaoka Y, Yoshida C, Fukuda T, Kajitani K, Ishiko O. Transcervical microwave myolysis for uterine myomas assisted by transvaginal ultrasonic guidance. J Obstet Gynaecol Res. 2009 Feb;35(1):145-51. doi: 10.1111/j.1447-0756.2008.00872.x. PMID 19215562
- [Background] Zhang J, Feng L, Zhang B, Ren J, Li Z, Hu D, Jiang X. Ultrasound-guided percutaneous microwave ablation for symptomatic uterine fibroid treatment--a clinical study. Int J Hyperthermia. 2011;27(5):510-6. doi: 10.3109/02656736.2011.562872. PMID 21756048
- [Background] Wang F, Zhang J, Han ZY, Cheng ZG, Zhou HY, Feng L, Hu DM. Imaging manifestation of conventional and contrast-enhanced ultrasonography in percutaneous microwave ablation for the treatment of uterine fibroids. Eur J Radiol. 2012 Nov;81(11):2947-52. doi: 10.1016/j.ejrad.2011.12.037. Epub 2012 Feb 16. PMID 22341698
- [Background] Yang Y, Zhang J, Han ZY, Yu MA, Ma X, Zhou HY, Hao YL, Zhao L, Dong XJ, Ge HL. Ultrasound-guided percutaneous microwave ablation for submucosal uterine fibroids. J Minim Invasive Gynecol. 2014 May-Jun;21(3):436-41. doi: 10.1016/j.jmig.2013.11.012. Epub 2013 Dec 4. PMID 24316137
- [Background] Zhao WP, Han ZY, Zhang J, Liang P. A retrospective comparison of microwave ablation and high intensity focused ultrasound for treating symptomatic uterine fibroids. Eur J Radiol. 2015 Mar;84(3):413-417. doi: 10.1016/j.ejrad.2014.11.041. Epub 2014 Dec 15. PMID 25572326
- [Background] Kanaoka Y, Hirai K, Ishiko O. Microwave endometrial ablation for menorrhagia caused by large submucous myomas. J Obstet Gynaecol Res. 2005 Dec;31(6):565-70. doi: 10.1111/j.1447-0756.2005.00338.x. PMID 16343261
- [Background] Reid PC, Coker A, Coltart R. Assessment of menstrual blood loss using a pictorial chart: a validation study. BJOG. 2000 Mar;107(3):320-2. doi: 10.1111/j.1471-0528.2000.tb13225.x. PMID 10740326
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Harding G, Coyne KS, Thompson CL, Spies JB. The responsiveness of the uterine fibroid symptom and health-related quality of life questionnaire (UFS-QOL). Health Qual Life Outcomes. 2008 Nov 12;6:99. doi: 10.1186/1477-7525-6-99. PMID 19014505
- [Derived] Jonsdottir G, Beermann M, Lundgren Cronsioe A, Hasselrot K, Kopp Kallner H. Ultrasound guided microwave ablation compared to uterine artery embolization treatment for uterine fibroids - a randomized controlled trial. Int J Hyperthermia. 2022;39(1):341-347. doi: 10.1080/02656736.2022.2034991. PMID 35134317